CLINICAL TRIAL: NCT01016392
Title: Kuvan® Adult Maternal Pediatric European Registry
Brief Title: Observational Study on the Long Term Safety of Kuvan® Treatment in Patients With Hyperphenylalaninemia (HPA) Due to Phenylketonuria (PKU) or BH4 Deficiency
Acronym: KAMPER
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR700773-001
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Hyperphenylalaninemia (HPA) Due to Phenylketonuria (PKU) or Tetrahydrobiopterin (BH4) Deficiency
Keywords: Observational post-authorization safety study on Kuvan®.
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Kuvan® is a synthetic copy of a body's own substance called tetrahydrobiopterin (BH4). BH4 is required by the body to use an amino acid called phenylalanine in order to build another substance called tyrosine.

Kuvan® received marketed authorisation in Europe in December 2008 and is now available in several European countries for the treatment of Hyperphenylalaninemia (HPA).

The primary objective is to assess the long-term safety in subjects treated with Kuvan®.

Secondary objectives are to provide additional information regarding:

* Safety in specific subject groups (elderly, pediatric, pregnant women and subjects with renal or hepatic insufficiency).
* Growth and neurocognitive outcomes for subjects with hyperphenylalaninemia (HPA) who are receiving treatment with Kuvan®.
* Progress and outcome of pregnancy for women with HPA who become pregnant while receiving treatment with Kuvan® (these women will be enrolled in a dedicated sub-registry).
* Assessment of adherence to diet and to Kuvan®.
* Assessment of long-term sensitivity to Kuvan®treatment.

DETAILED DESCRIPTION:
This is an observational, multicenter, drug registry Study. The study will have a total duration of 15 years, including a 10-year inclusion period. No diagnostic, therapeutic or experimental intervention is involved. Subjects will receive clinical assessments, medications and treatments solely as determined by their study physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult or pediatric subject (no age limit) of either gender with HPA due to PKU or BH4 deficiency.
* Have been shown to be responsive to BH4 or Kuvan. (Note: For Spain only-Have been shown to be responsive to BH4 or for the newly diagnosed subjects to be responsive to Kuvan as defined in the Summary of Product Characteristics [SmPC]).
* Currently being treated with Kuvan® at a participating centre.
* Subject or parent/legal guardian willing and able to provide written signed informed consent and given before any data collection. If a child is old enough to read and write, a separate assent form will be given.

Exclusion Criteria:

* Known hypersensitivity to Kuvan®
* Legal incapacity or limited legal capacity without legal guardian representation
* Breast-feeding

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with HPA due to PKU or BH4 deficiency followed at participating centres.
  And specific groups (elderly, pediatric, pregnant women and subjects with renal or hepatic insufficiency).
Sampling Method: Non-Probability Sample
Enrollment: 627 (Actual)
Dates: Start 2009-12; Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence and description of Adverse Events and Serious Adverse Events (AEs/SAEs) | A maximum of 15 years treatment duration.

SECONDARY OUTCOMES:
Incidence of AEs/SAEs in specific population (elderly, children, subjects with renal or hepatic insufficiency) | A maximum of 15 years treatment duration.
Description on somatic growth (in BH4 deficient children < 3 years) | A maximum of 15 years treatment duration.
Neurocognitive outcomes | A maximum of 15 years treatment duration.
Neurological and psychiatric assessment | A maximum of 15 years treatment duration.
Diet and Kuvan® treatment adherence | A maximum of 15 years treatment duration.
Long-term sensitivity to Kuvan® treatment | A maximum of 15 years treatment duration.
Blood Phe levels | A maximum of 15 years treatment duration.
Tyrosine (Tyr) levels | A maximum of 15 years treatment duration.
Pregnancy and delivery outcomes | A maximum of 15 years treatment duration.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Kucuksayrac, MD, Study Director — BioMarin Pharmaceutical
Locations (69):
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
- France (21):
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site - Armand Trousseau, Paris
  - Research Site - Necker, Paris
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Tarbes
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
- Germany (12):
  - Research Site, Berlin
  - Research Site, Cottbus
  - Research Site, Düsseldorf
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, München
  - Research Site, Münster
  - Research Site, Reutlingen
- Italy (9):
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Genova
  - Research Site, Milan
  - Research Site - Ospedale Annunziata, Napoli
  - Research Site - Policlinico Federico, Napoli
  - Research Site, Padua
  - Research Site, Roma
- Netherlands (5):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Maastricht
  - Research Site, Rotterdam
  - Research Site, Utrecht
- Research Site, Porto, Portugal
- Slovakia (2):
  - Research Site, Banská Bystrica
  - Research Site, Košice
- Spain (12):
  - Research Site, Bilbao
  - Research Site, Esplugues de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Santander
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Zaragoza
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Stockholm
  - Research Site, Uppsala